CLINICAL TRIAL: NCT04157751
Title: A Multicentre, Randomised, Double-blind, 90-day Superiority Trial to Evaluate the Effect on Clinical Benefit, Safety and Tolerability of Once Daily Oral EMPagliflozin 10 mg Compared to Placebo, Initiated in Patients Hospitalised for acUte Heart faiLure (de Novo or Decompensated Chronic HF) Who Have Been StabilisEd (EMPULSE)
Brief Title: A Study to Test the Effect of Empagliflozin in Patients Who Are in Hospital for Acute Heart Failure
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1245-0204; 2019-002946-19 (EudraCT Number)
Record Dates: First submitted 2019-11-04; First posted 2019-11-08 (Actual); Results first posted 2022-06-06 (Actual); Last update posted 2022-07-19 (Actual); Status verified 2022-06

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure | interventions — empagliflozin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Empagliflozin (Experimental)
  Interventions: Drug: Empagliflozin
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo to Empagliflozin

INTERVENTIONS:
Drug: Empagliflozin — Film-coated tablet
  Arms: Empagliflozin
Drug: Placebo to Empagliflozin — Film-coated tablet
  Arms: Placebo

SUMMARY:
This is a study in adults who are in hospital for acute heart failure. The purpose of this study is to find out whether starting to take a medicine called empagliflozin soon after first being treated in hospital helps people with acute heart failure.

Participants are in the study for about 3 months. At the beginning, participants are still in hospital. Later, they visit the hospital about 3 times and get 1 phone call. Participants are put into 2 groups by chance. One group takes 1 empagliflozin tablet a day. The other group takes

1 placebo tablet a day. Placebo tablets look like empagliflozin tablets but do not contain any medicine. Empagliflozin belongs to a class of medicines known as SGLT-2 inhibitors. It is used to treat type 2 diabetes.

During the study, the doctors check whether participants have additional heart failure events like needing to go to the hospital again because of heart failure. The participants answer questions about how their heart failure affects their life. We then compare the results between the empagliflozin and placebo groups. The doctors also regularly check the general health of the participants.

ELIGIBILITY:
Inclusion Criteria:

* Currently hospitalised for the primary diagnosis of acute heart failure (de novo or decompensated chronic HF), regardless of ejection fraction (EF). Patients with a diagnosis of hospitalized heart failure must have HF symptoms at the time of hospital admission
* Evidence of left ventricular ejection fraction (LVEF, either reduced or preserved EF) as per local reading preferably measured during current hospitalisation or in the 12 months prior to randomisation
* Patients must be randomised after at least 24 hours and no later than 5 days after admission, as early as possible after stabilization and while still in hospital
* Patients must fulfil the following stabilisation criteria (while in the hospital):

  * SBP ≥100mm Hg and no symptoms of hypotension in the preceding 6 hours,
  * no increase in i.v. diuretic dose for 6 hours prior to randomisation,
  * no i.v. vasodilators including nitrates within the last 6 hours prior to randomisation
  * no i.v. inotropic drugs for 24 hours prior to randomisation.
* Elevated NT-proBNP ≥ 1600pg/mL or BNP ≥400 pg/mL according to the local lab, for patients without atrial fibrillation (AF); or elevated NT-proBNP ≥ 2400pg/mL or BNP ≥600 pg/mL for patients with AF, measured during the current hospitalization or in the 72 hours prior to hospital admission,. For patients treated with an angiotensin receptor neprilysin inhibitor (ARNI) in the previous 4 weeks prior to randomisation, only NT-proBNP values should be used
* HF episode leading to hospitalisation must have been treated with a minimum single dose of 40 mg of i.v. furosemide (or equivalent i.v. loop diuretic defined as 20 mg of torasemide or 1 mg of bumetanide)
* Further Inclusion Criteria Apply

Exclusion Criteria:

* Cardiogenic shock
* Current hospitalisation for acute heart failure primarily triggered by pulmonary embolism, cerebrovascular accident, or acute myocardial infarction (AMI)
* Current hospitalisation for acute heart failure not caused primarily by intravascular volume overload;
* Below interventions in the past 30 days prior to randomisation or planned during the study:

  * Major cardiac surgery, or TAVI (Transcatheter Aortic Valve Implantation), or PCI, or Mitraclip
  * All other surgeries that are considered major according to investigator judgement
  * Implantation of cardiac resynchronisation therapy (CRT) device
  * cardiac mechanical support implantation
  * Carotid artery disease revascularisation (stent or surgery)
* Acute coronary syndrome / myocardial infarction, stroke or transient ischemic attack (TIA) in the past 90 days prior to randomisation
* Heart transplant recipient, or listed for heart transplant with expectation to receive a transplant during the course of this trial (according to investigator judgement), or planned for palliative care for HF, or currently using left ventricular assist device (LVAD) or intra-aortic balloon pump (IABP) or any other type of mechanical circulatory support, or patients on mechanical ventilation, or patients with planned inotropic support in an outpatient setting
* Haemodynamically significant (severe) uncorrected primary cardiac valvular disease planned for surgery or intervention during the course of the study (note: secondary mitral regurgitation or tricuspid regurgitation due to dilated cardiomyopathy is not excluded unless planned for surgery or intervention during the course of the study)
* Impaired renal function, defined as eGFR < 20 mL/min/1.73 m2 as measured during hospitalization (latest local lab measurement before randomisation) or requiring dialysis
* Type 1 Diabetes Mellitus (T1DM)
* History of ketoacidosis, including diabetic ketoacidosis (DKA)
* Further Exclusion Criteria Apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 530 (Actual)
Dates: Start 2020-05-18 (Actual); Primary Completion 2021-05-28 (Actual); Study Completion 2021-06-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (118):
- United States (30):
  - University of Southern California, Los Angeles, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - University of California Irvine, Orange, California
  - The Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center, Torrance, California
  - Cardiology Associates Research Co., Daytona Beach, Florida
  - University of Florida Health Jacksonville, Jacksonville, Florida
  - Grady Memorial Hospital, Atlanta, Georgia
  - Methodist Medical Center, Peoria, Illinois
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - United Hospital, Saint Paul, Minnesota
  - University Of Mississippi Medical Center, Jackson, Mississippi
  - Saint Luke's Hospital of Kansas City, Kansas City, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Cardiovascular Associates of the Delaware Valley, Elmer, New Jersey
  - Jefferson Washington Township Hospital, Washington Township, New Jersey
  - Erie County Medical Center, Buffalo, New York
  - The DeMatteis Center for Cardiac Research and Education, Greenvale, New York
  - Stony Brook Medicine, Stony Brook, New York
  - Montefiore Medical Center, The Bronx, New York
  - The University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - North Carolina Heart and Vascular, Raleigh, North Carolina
  - University of Oklahoma, Oklahoma City, Oklahoma
  - South Oklahoma Heart Research Group, Oklahoma City, Oklahoma
  - Ralph H. Johnson VA Medical Center, Charleston, South Carolina
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Pharmatex Research, Amarillo, Texas
  - Center for Advanced Cardiac Care - Heart Failure Clinic, Plano, Texas
  - Inova Fairfax Medical Campus, Falls Church, Virginia
  - Sentara Norfolk General Hospital, Norfolk, Virginia
  - University of Wisconsin, Madison, Wisconsin
- Belgium (7):
  - Aalst - HOSP Onze-Lieve-Vrouw, Aalst
  - Brussels - UNIV UZ Brussel, Brussels
  - AZ Sint-Blasius, Dendermonde
  - Ziekenhuis Oost-Limburg - Campus Sint-Jan, Genk
  - UZ Leuven, Leuven
  - Liège - HOSP CHR de la Citadelle, Liège
  - UNIV Ambroise Paré, Mons
- Canada (3):
  - Royal Jubilee Hospital, Victoria, British Columbia
  - St. Boniface General Hospital, Winnipeg, Manitoba
  - Toronto General Hospital, Toronto, Ontario
- China (6):
  - Beijing Chao-Yang Hospital, Beijing
  - Beijing AnZhen Hospital, Beijing
  - The First Hospital of Jilin University, Changchun
  - West China Hospital, Chengdu
  - First Affiliated Hospital of Xi'an JiaoTong University, Xi'an
  - Xiamen Cardiovascular Hospital Xiamen University, Xiamen
- Czechia (4):
  - University Hospital Brno, Brno
  - Univ.Hosp U Svate Anny, I.Internal Clinic-Cardiology,Brno, Brno
  - University Hospital Motol, Prague
  - District Hospital, Tabor, Tábor
- Denmark (5):
  - Aalborg Universitetsshospital, Aalborg
  - Frederiksberg Hospital, Frederiksberg
  - Herlev and Gentofte Hospital, Herlev
  - Hvidovre Hospital, Hvidovre
  - Viborg Regionhospital, Viborg
- Germany (11):
  - Charité - Universitätsmedizin Berlin, Berlin
  - Bremer Institut für Herz- und Kreislaufforschung (BIHKF) am Klinikum Links der Weser, Bremen
  - Herzzentrum Dresden GmbH Universitätsklinik, Dresden
  - Universitäts-Herzzentrum Freiburg, Bad Krozingen GmbH, Freiburg im Breisgau
  - Universitätsklinikum Gießen und Marburg GmbH, Giessen
  - Universitätsklinikum Jena, Jena
  - Asklepios Klinik Langen-Seligenstadt GmbH, Langen
  - Klinikum Leverkusen gGmbH, Leverkusen, Leverkusen
  - Klinikum der Stadt Ludwigshafen am Rhein gGmbH, Ludwigshafen
  - Universitätsklinikum Schleswig-Holstein, Campus Lübeck, Lübeck
  - Universitätsklinikum Würzburg AÖR, Würzburg
- Hungary (5):
  - Semmelweis University, Budapest
  - University Debrecen Hospital, Debrecen
  - University of Pecs, Pécs
  - Csongrad Country Dr Bugyi Istvan Hosp., Szentes
  - Fejer County Saint George University Teaching Hospital, Székesfehérvár
- Italy (10):
  - ASST degli Spedali Civili di Brescia, Brescia
  - Università degli Studi "Magna Grecia" - Campus "S. Venuta", Catanzaro
  - Ospedale della Val di Chiana Santa Margherita, Cortona
  - Az.Osp. Universitaria "Ospedali Riuniti", Foggia
  - Centro Cardiologico Monzino-IRCCS, Milan
  - ASST Grande Ospedale Metropolitano Niguarda, Milan
  - Osp. Guglielmo da Saliceto AUSL di Piacenza, Piacenza
  - IRCCS San Raffaele, Roma
  - AO Città della Salute e della, Torino
  - Azienda Sanitaria Universitaria Giuliano Isontina, Trieste
- Japan (9):
  - Japan Community Health Care Organization Kyushu Hospital, Fukuoka, Kitakyushu
  - Mito Medical Center, Ibaraki, Higashiibaraki-gun
  - Kanagawa Cardiovascular and Respiratory Center, Kanagawa, Yokohama
  - Shinshu University Hospital, Nagano, Matsumoto
  - The Sakakibara Heart Institute of Okayama, Okayama, Okayama
  - Osaka University Hospital, Osaka, Suita
  - Kawaguchi Cardiovascular and Respiratory Hospital, Saitama, Kawaguchi
  - Saitama Sekishikai Hospital, Saitama, Sayama
  - Nihon University Itabashi Hospital, Tokyo, Itabashi-ku
- Netherlands (10):
  - Jeroen Bosch Ziekenhuis-Hertogenbosch, 's-Hertogenbosch
  - Gelre Ziekenhuizen Apeldoorn, Apeldoorn
  - TREANT Zorggroep, Emmen
  - Groene Hart ziekenhuis, Gouda
  - Universitair Medisch Centrum Groningen, Groningen
  - Sint Jansdal Ziekenhuis, Harderwijk
  - Alrijne Leiderdorp, Leiderdorp
  - Bravis ziekenhuis, locatie Roosendaal, Roosendaal
  - HagaZiekenhuis, The Hague
  - Diakonessenhuis Utrecht, Utrecht
- Norway (5):
  - Helse Førde HF, Førde Sentralsjukehus, Førde
  - Sykehuset Innlandet HF, Avd. Lillehammer, Lillehammer
  - Akershus Universitetssykehus HF, Lørenskog
  - Helse Stavanger, Stavanger Universitetssykehus, Stavanger
  - Universitetssykehuset Nord-Norge, Tromsø, Tromsø
- Poland (4):
  - Saint Wincenty a Paulo Hosp., Cardiology Dept., Gdynia, Gdynia
  - Card.Cli.Mil.Med.Ac.Uni.Cli.Hosp. Cent.Vetera.Hosp.Lodz, Lodz
  - Cent.Clin.Hosp.Med.Univ.Lodz,Electrocard, Lodz
  - Provincial Specialist M. Kopernik Hospital, Lodz
- Spain (7):
  - Hospital Universitario Virgen de la Arrixaca, El Palmar
  - Hospital de Bellvitge, L'Hospitalet de Llobregat
  - Hospital Puerta de Hierro, Majadahonda
  - Hospital Virgen de la Victoria, Málaga
  - Hospital Moises Broggi, Sant Joan Despí
  - Hospital Nuestra Señora de Valme, Seville
  - Hospital Clínico de Valencia, Valencia
- Sweden (2):
  - Sahlgrenska US, Göteborg, Gothenburg
  - Sahlgrenska Universitetssjukhuset, Östra, Gothenburg

IPD SHARING:
Plan to Share IPD: Yes
After the study is completed and the primary manuscript is accepted for publishing, researchers can use this following link https://www.mystudywindow.com/msw/datasharing to request access to the clinical study documents regarding this study, and upon a signed "Document Sharing Agreement".
  Also, Researchers can use the following link https://www.mystudywindow.com/msw/datasharing to find information in order to request access to the clinical study data, for this and other listed studies, after the submission of a research proposal and according to the terms outlined in the website.
  The data shared are the raw clinical study data sets.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: After all regulatory activities are completed in the US and EU for the product and indication, and after the primary manuscript has been accepted for publication.
Access Criteria: For study documents - upon signing of a 'Document Sharing Agreement'. For study data - 1. after the submission and approval of the research proposal (checks will be performed by both the independent review panel and the sponsor, including checking that the planned analysis does not compete with sponsor's publication plan); 2. and upon signing of a 'Data Sharing Agreement'.
URL: https://www.mystudywindow.com/msw/datasharing

REFERENCES:
- [Derived] Jongs N, Gasparyan SB, Frison L, Schloemer P, Brinker M, Little DJ, Heerspink HJL. Use of eGFR Slope Thresholds as End Point Components in a Kidney Disease Progression Hierarchical Composite End Point. J Am Soc Nephrol. 2025 Dec 1;36(12):2421-2430. doi: 10.1681/ASN.0000000766. Epub 2025 Jun 17. PMID 40526444
- [Derived] Ferreira JP, Blatchford JP, Teerlink JR, Kosiborod MN, Angermann CE, Biegus J, Collins SP, Tromp J, Nassif ME, Psotka MA, Comin-Colet J, Mentz RJ, Brueckmann M, Nordaby M, Ponikowski P, Voors AA. Mineralocorticoid receptor antagonist use and the effects of empagliflozin on clinical outcomes in patients admitted for acute heart failure: Findings from EMPULSE. Eur J Heart Fail. 2023 Oct;25(10):1797-1805. doi: 10.1002/ejhf.2982. Epub 2023 Aug 22. PMID 37540060
- [Derived] Kosiborod MN, Angermann CE, Collins SP, Teerlink JR, Ponikowski P, Biegus J, Comin-Colet J, Ferreira JP, Mentz RJ, Nassif ME, Psotka MA, Tromp J, Brueckmann M, Blatchford JP, Salsali A, Voors AA. Effects of Empagliflozin on Symptoms, Physical Limitations, and Quality of Life in Patients Hospitalized for Acute Heart Failure: Results From the EMPULSE Trial. Circulation. 2022 Jul 26;146(4):279-288. doi: 10.1161/CIRCULATIONAHA.122.059725. Epub 2022 Apr 4. PMID 35377706
- [Derived] Voors AA, Angermann CE, Teerlink JR, Collins SP, Kosiborod M, Biegus J, Ferreira JP, Nassif ME, Psotka MA, Tromp J, Borleffs CJW, Ma C, Comin-Colet J, Fu M, Janssens SP, Kiss RG, Mentz RJ, Sakata Y, Schirmer H, Schou M, Schulze PC, Spinarova L, Volterrani M, Wranicz JK, Zeymer U, Zieroth S, Brueckmann M, Blatchford JP, Salsali A, Ponikowski P. The SGLT2 inhibitor empagliflozin in patients hospitalized for acute heart failure: a multinational randomized trial. Nat Med. 2022 Mar;28(3):568-574. doi: 10.1038/s41591-021-01659-1. Epub 2022 Feb 28. PMID 35228754
- See also: Related Info — http://www.mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A multicentre, randomised, double-blind trial to assess whether in-hospital administration of empagliflozin results in improvement in heart failure-related outcomes compared to placebo in patients with acute heart failure.
Pre-assignment Details: All subjects were screened for eligibility prior to participation in the trial. Subjects attended a specialist site which ensured that they (the subjects) strictly met all inclusion and none of the exclusion criteria. Subjects were not to be allocated to a treatment group if any of the entry criteria were violated.
Groups:
- Placebo: 1 film-coated tablet of placebo matching 10 mg empagliflozin was administered orally once daily in patients with acute heart failure.
- 10 mg Empagliflozin: 1 film-coated tablet of 10 milligram (mg) of empagliflozin was administered orally once daily in patients with acute heart failure.
Period: Overall Study
Arm/Group | Placebo | 10 mg Empagliflozin
Started (Randomised) | 265 | 265
Treated | 264 | 260
Completed | 202 | 208
Not Completed | 63 | 57
Not completed — Withdrawal by Subject | 12 | 17
Not completed — Lost to Follow-up | 6 | 2
Not completed — Adverse Event | 34 | 23
Not completed — Not treated | 1 | 5
Not completed — Other reason not stated above | 10 | 10

BASELINE CHARACTERISTICS:
Population: Randomised Set (RS), including all randomised patients.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | 10 mg Empagliflozin | Total
Number analyzed (Participants) | 265 | 265 | 530
Age, Continuous [Mean (Standard Deviation); unit: Years] | 68.1 (13.8) | 68.9 (12.6) | 68.5 (13.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 93 | 86 | 179
  Male | 172 | 179 | 351
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9 | 6 | 15
  Not Hispanic or Latino | 256 | 259 | 515
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 0 | 2
  Asian | 25 | 32 | 57
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 33 | 21 | 54
  White | 202 | 211 | 413
  More than one race | 2 | 1 | 3
  Unknown or Not Reported | 1 | 0 | 1
Kansas City cardiomyopathy questionnaire-Total symptom score (KCCQ-TSS) [Mean (Standard Deviation); unit: Score on a scale] — The Kansas City Cardiomyopathy Questionnaire is a self-administered questionnaire that includes 23 items that map to 7 domains: symptom frequency, symptom burden, symptom stability, physical limitations, social limitations, quality of life and self-efficacy. The symptom frequency and symptom burden domains are merged into a total symptom score. Scores are represented on a 0-to-100-point scale, where a higher score reflects a better health status. KCCQ-TSS at baseline is reported. Only participants in the randomised set and with non-missing data are included. Population: Only participants in the randomised set and with non-missing data are included.
  Score on a scale
    number analyzed (Participants) | 264 | 262 | 526
    (all) | 41.91 (23.98) | 39.71 (24.06) | 40.81 (24.02)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Pairwise Comparisons With Wins of Clinical Benefit, a Composite of Death, Number of Heart Failure Events (HFEs), Time to the First HFE and ≥5-point Difference in CfB in KCCQ-TSS After 90 Days of Treatment
Description: Clinical benefit, a composite of death, number of HFEs, time to first HFE and change from baseline (CfB) in Kansas City Cardiomyopathy Questionnaire-Total Symptom Score (KCCQ-TSS) after 90 days of treatment. All patients randomised to empagliflozin are compared to all patients randomised to placebo within strata. For any two patients, a patient will win, i.e. achieve a better clinical outcome, as determined by assessing the following criteria sequentially, stopping when an advantage for either patient is shown:
  1. Death: death is worse than no death; earlier death is worse; tied if not possible to determine.
  2. Number of HFEs: more HFEs is worse; tied, if same number of HFEs.
  3. Time to first HFE: earlier HFE is worse; tied, if not possible to determine.
  4. KCCQ-TSS CfB at Day 90: more positive CfB is better; the threshold for the difference is >= 5 for a win; tied, if difference < 5.
  The KCCQ-TSS ranges from 0 to 100, where a higher score reflects a better outcome.
  pct. = percentage
Time Frame: Up to 90 days. For KCCQ-TSS: at baseline and at day 90.
Population: Randomised Set (RS), including all randomised patients.
Measure: Number; unit: pct. (%) of winning pairwise comparisons
Units Other Than Participants: Pairwise comparisons
Arm/Group | Placebo | 10 mg Empagliflozin
Number analyzed (Participants) | 265 | 265
Number analyzed (Pairwise comparisons) | 39162 | 39162
pct. (%) of winning pairwise comparisons
  Time to death | 4.01 | 7.15
  Frequency of HFEs | 7.65 | 10.59
  Time to HFE | 0.57 | 0.24
  KCCQ-TSS change from baseline (>=5-point difference) | 27.48 | 35.91
Statistical Analysis 1: Comparison: Placebo vs 10 mg Empagliflozin; Stratified win ratio (WR) was used, calculated as total number of wins in the empa group across all strata divided by total number of losses. Weights were applied analogous to a Mantel-Haenszel approach. 1. death in pbo first; 2. death in empa first; 3. HFEs in pbo more frequently; 4. HFEs in empa more frequently; 5. HFEs in pbo first; 6. HFEs in empa first; 7. KCCQ-TSS change lower in pbo; 8. KCCQ-TSS change lower in empa; Test type: Other; p = 0.0027, Asymptotic normal U statistics approach — p-value for WR<=1.0 (one-sided), variance calculated using the asymptotic normal U statistics approach; Stratified Win Ratio = 1.36, 95% CI 2-sided [1.09 to 1.68] — WR estimate= [((a)+(c)+(e)+(g)) / ((b)+(d)+(f)+(h))]

2. Secondary Outcome: Number of Participants With Improvement of at Least 10 Points in KCCQ-TSS After 90 Days of Treatment
Description: Number of participants with improvement of at least 10 points in Kansas City Cardiomyopathy Questionnaire - Total Symptom Score (KCCQ-TSS) from baseline after 90 days of treatment.
  The Kansas City Cardiomyopathy Questionnaire is a self-administered questionnaire that includes 23 items that map to 7 domains: symptom frequency, symptom burden, symptom stability, physical limitations, social limitations, quality of life and self-efficacy. The symptom frequency and symptom burden domains are merged into the total symptom score. Scores are represented on a 0-to-100-point scale, where a higher score reflects a better health status.
Time Frame: At baseline and at day 90.
Population: Randomised Set (RS), including all randomised patients.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | 10 mg Empagliflozin
Number analyzed (Participants) | 265 | 265
Participants | 202 | 220
Statistical Analysis 1: Comparison: Placebo vs 10 mg Empagliflozin; Logistic regression including terms for baseline KCCQ-TSS, treatment and heart failure status; Test type: Other; p = 0.0970, Regression, Logistic — p-value for OR=1.0 (two-sided); Wald Confidence interval; Odds Ratio (OR) = 1.522, 95% CI 2-sided [0.927 to 2.501], Standard Error of Mean 0.386 — Comparison vs. Placebo

3. Secondary Outcome: Change From Baseline in KCCQ-TSS After 90 Days of Treatment
Description: Change from baseline in Kansas City Cardiomyopathy Questionnaire - Total Symptom Score (KCCQ-TSS).
  The Kansas City Cardiomyopathy Questionnaire is a self-administered questionnaire that includes 23 items that map to 7 domains: symptom frequency, symptom burden, symptom stability, physical limitations, social limitations, quality of life and self-efficacy. The symptom frequency and symptom burden domains are merged into the total symptom score. The score is represented on a 0-to-100-point scale, where a higher score reflects a better health status.
  Change from baseline in KCCQ-TSS at day 90 was modeled using a MMRM with visit (day 15 and day 30) as repeated measures, adjusted mean (standard error) after 90 days of treatment is reported.
Time Frame: At baseline, at day 15, 30 and at day 90.
Population: Patients in the randomised set (RS) and with non-missing data for this endpoint. Observed case including data after treatment discontinuation (OC-AD).
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Placebo | 10 mg Empagliflozin
Number analyzed (Participants) | 221 | 230
Score on a scale | 31.73 (1.49) | 36.19 (1.48)
Statistical Analysis 1: Comparison: Placebo vs 10 mg Empagliflozin; Restricted maximum likelihood estimation based on a mixed-effect model for repeated measures (MMRM) analysis to obtain adjusted means for the treatment effects. This model included discrete fixed effects for treatment group, and heart failure status at each visit and continuous fixed effects for baseline value at each visit. Missing data caused by patient withdrawal or other reasons were handled implicitly by the MMRM approach. Unstructured covariance structure was used; Test type: Other; p = 0.0347, Mixed Models Analysis — p-value for difference = 0 (two-sided); Difference of adjusted mean = 4.45, 95% CI 2-sided [0.32 to 8.59], Standard Error of Mean 2.10

4. Secondary Outcome: Change From Baseline in Log-transformed N-Terminal Pro-Brain Natriuretic Peptide (NTproBNP) Area Under the Curve (AUC) Over 30 Days of Treatment
Description: Change from baseline in log-transformed N-Terminal Pro-Brain Natriuretic Peptide (NTproBNP) Area under the curve (AUC) over 30 days of treatment is reported.
Time Frame: From baseline to day 30.
Population: Patients included the randomised set (RS), and with non-missing data for this endpoint.
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: Picogram/milliliter * days
Arm/Group | Placebo | 10 mg Empagliflozin
Number analyzed (Participants) | 256 | 255
Picogram/milliliter * days | 26.77 [25.15 to 28.48] | 24.07 [22.61 to 25.62]
Statistical Analysis 1: Comparison: Placebo vs 10 mg Empagliflozin; Area under the curve (AUC) of change from baseline in log-transformed NT-proBNP level over 30 days of treatment was analysed by an analysis of covariance (ANCOVA). NT-proBNP level is regarded as log-normally distributed, therefore values were log-transformed prior to analysis. The linear trapezoidal rule was used to calculate the AUC after the log-transformation had been applied to each value; Test type: Other; p = 0.0176, ANCOVA; ANCOVA with a discrete fixed effect for heart failure status and a continuous fixed effect for baseline NT-proBNP level; Adjusted geometric mean ratio = 0.90, 95% CI 2-sided [0.82 to 0.98] — Comparison vs. Placebo

5. Secondary Outcome: Percentage of Days Alive and Out of Hospital (DAOH) From Study Drug Initiation Until 30 Days After Initial Hospital Discharge
Description: The follow-up time for DAOH analyses was defined as 30 days after initial hospital discharge, or time between initial hospital discharge and date of censoring for non-fatal events except for patients who died within the first 30 days, where 30 days was considered as the DAOH follow-up time.
  DAOH for each patient was calculated as follow-up time subtracted by the number of days in hospital during the 30 days after initial hospital discharge as well as the number of days being dead within the 30 days. Percentage DAOH was defined as DAOH divided by the DAOH follow-up time of each patient multiplied by 100.
Time Frame: Up to 30 days after initial hospital discharge.
Population: Patients included the treated set (TS), and with non-missing data for this endpoint. TS includes all patients treated with at least one dose of trial medication.
Measure: Mean (Standard Deviation); unit: DAOH in percentage (%)
Arm/Group | Placebo | 10 mg Empagliflozin
Number analyzed (Participants) | 264 | 258
DAOH in percentage (%) | 80.90 (21.25) | 81.37 (18.62)

6. Secondary Outcome: Percentage of Days Alive and Out of Hospital (DAOH) From Study Drug Initiation Until 90 Days After Randomisation
Description: The follow-up time for DAOH analyses was defined as 90 days after randomisation, or time between randomisation and date of censoring for non-fatal events except for patients who died within the first 90 days, where 90 days was considered as the DAOH follow-up time. DAOH for each patient was calculated as follow-up time subtracted by the number of days in hospital during the 90 days after randomisation as well as the number of days being dead within the first 90 days.
  Percentage DAOH was defined as DAOH divided by the DAOH follow-up time of each patient multiplied by 100.
Time Frame: Up to 90 days after randomisation.
Population: Patients in the treated set (TS) and with non-missing data for this endpoint.
Measure: Mean (Standard Deviation); unit: DAOH in percentage (%)
Arm/Group | Placebo | 10 mg Empagliflozin
Number analyzed (Participants) | 260 | 257
DAOH in percentage (%) | 85.79 (22.76) | 87.55 (19.54)

7. Secondary Outcome: Incidence Rate of First Occurrence of Cardiovascular (CV) Death or Heart Failure Event (HFE) Until End of Trial Visit
Description: Incidence rate of first occurrence of CV death or HFE until end of trial visit per 100 patient-year (pt-yrs) at risk is reported.
  Incidence rate per 100 pt-yrs = 100* number of patients with event / time at risk [years].
Time Frame: Up to 127 days.
Population: Randomised Set (RS), including all randomised patients.
Measure: Number (95% Confidence Interval); unit: Patients with events / 100pt-yrs at risk
Arm/Group | Placebo | 10 mg Empagliflozin
Number analyzed (Participants) | 265 | 265
Patients with events / 100pt-yrs at risk | 78.81 [58.11 to 102.62] | 55.01 [38.10 to 74.99]
Statistical Analysis 1: Comparison: Placebo vs 10 mg Empagliflozin; Test type: Other; p = 0.1241, Regression, Cox — p-value for HR=1.0 (two sided); Cox proportional hazard model with terms for heart failure status and treatment; Hazard Ratio (HR) = 0.71, 95% CI 2-sided [0.46 to 1.10] — Comparison vs. Placebo

8. Secondary Outcome: Number of Participants With Hospitalization for Heart Failure (HHF) Until 30 Days After Initial Hospital Discharge
Description: Number of participants with hospitalization for heart failure (HHF) until 30 days after initial hospital discharge.
Time Frame: Up to 30 days after initial hospital discharge.
Population: Randomised Set (RS), including all randomised patients.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | 10 mg Empagliflozin
Number analyzed (Participants) | 265 | 265
Participants | 12 | 14

9. Secondary Outcome: Composite Renal Endpoint: Number of Participants With Chronic Dialysis, Renal Transplant, Sustained Reduction in eGFR(CKD-EPI)cr
Description: The occurrence of the composite renal endpoint:
  * chronic dialysis (with a frequency of twice per week or more for at least 90 days), or
  * renal transplant, or
  * sustained reduction in Glomerular filtration rate estimated by the chronic kidney disease epidemiology collaboration formula with serum creatinine measurement (eGFR (CKD-EPI)cr) from baseline of ≥40%, or
  * sustained eGFR [mL/min/1.73 m2] <15 and baseline value ≥30, or
  * sustained eGFR <10 and baseline value <30; is reported by number of participants with component events. (These events may have occurred after the endpoint was already met. Combinations may not have occurred on the same day).
  Sustained was determined by 2 or more consecutive post-baseline central laboratory measurements separated by at least 30 days.
Time Frame: Up to 90 days.
Population: Randomised Set (RS), including all randomised patients.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | 10 mg Empagliflozin
Number analyzed (Participants) | 265 | 265
Participants | 2 | 0

10. Secondary Outcome: Weight Change Per Mean Daily Loop Diuretic Dose After 15 Days of Treatment
Description: Diuretic effect as assessed by weight change per mean daily loop diuretic dose after 15 days of treatment.
  Diuretic dose = 40 mg intravenous furosemide or 80 mg oral furosemide.
  Abbreviation:
  Kg: Kilogram
Time Frame: At baseline and at day 15.
Population: Patients in the randomised set (RS) and with non-missing values for this endpoint.
Measure: Mean (Standard Deviation); unit: Kg per loop diuretic dose
Arm/Group | Placebo | 10 mg Empagliflozin
Number analyzed (Participants) | 224 | 212
Kg per loop diuretic dose | -2.43 (23.46) | -4.45 (16.65)

11. Secondary Outcome: Weight Change Per Mean Daily Loop Diuretic Dose After 30 Days of Treatment
Description: Diuretic effect as assessed by weight change per mean daily loop diuretic dose after 30 days of treatment.
  Diuretic dose = 40 mg intravenous furosemide or 80 mg oral furosemide
  Abbreviation:
  Kg: Kilogram
Time Frame: At baseline and at day 30.
Population: Patients in the randomised set (RS) and with non-missing values for this endpoint.
Measure: Mean (Standard Deviation); unit: Kg per loop diuretic dose
Arm/Group | Placebo | 10 mg Empagliflozin
Number analyzed (Participants) | 216 | 219
Kg per loop diuretic dose | -2.69 (21.74) | -6.91 (25.34)

ADVERSE EVENTS:
Time Frame: [All-cause Mortality]: From first study drug intake until end of follow-up, up to 202 days. [Serious and Other Adverse Event]: From first study drug intake until 7 days after last intake of study medication, up to 127 days.
Description: [All-cause Mortality]: Randomised Set (RS) including all randomised patients. [Serious and Other Adverse Events]: Treated Set (TS), consisting of all patients treated with at least once dose of trial medication.
Arm/Group | Placebo | 10 mg Empagliflozin
All-Cause Mortality (participants affected / at risk) | 22/265 | 11/265
Serious Adverse Events (participants affected / at risk) | 115/264 | 84/260
Other Adverse Events (participants affected / at risk) | 19/264 | 20/260
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=264) | 10 mg Empagliflozin (N=260)
Acute left ventricular failure (Cardiac disorders) | 2 | 0
Acute myocardial infarction (Cardiac disorders) | 1 | 0
Aortic valve incompetence (Cardiac disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 2 | 3
Atrial flutter (Cardiac disorders) | 2 | 1
Atrial thrombosis (Cardiac disorders) | 1 | 1
Bradycardia (Cardiac disorders) | 0 | 3
Cardiac arrest (Cardiac disorders) | 5 | 2
Cardiac failure (Cardiac disorders) | 37 | 25
Cardiac failure acute (Cardiac disorders) | 3 | 3
Cardiac failure chronic (Cardiac disorders) | 2 | 2
Cardiac failure congestive (Cardiac disorders) | 11 | 2
Cardiac ventricular thrombosis (Cardiac disorders) | 0 | 1
Cardiogenic shock (Cardiac disorders) | 1 | 1
Chronic left ventricular failure (Cardiac disorders) | 3 | 1
Coronary artery disease (Cardiac disorders) | 0 | 2
Coronary artery occlusion (Cardiac disorders) | 2 | 0
Coronary artery stenosis (Cardiac disorders) | 0 | 2
Coronary ostial stenosis (Cardiac disorders) | 1 | 0
Mitral valve incompetence (Cardiac disorders) | 1 | 1
Myocardial infarction (Cardiac disorders) | 3 | 0
Myocardial ischaemia (Cardiac disorders) | 0 | 1
Silent myocardial infarction (Cardiac disorders) | 1 | 0
Sinus node dysfunction (Cardiac disorders) | 1 | 1
Ventricular arrhythmia (Cardiac disorders) | 1 | 0
Ventricular fibrillation (Cardiac disorders) | 1 | 0
Ventricular tachycardia (Cardiac disorders) | 7 | 8
Gastrointestinal arteriovenous malformation (Congenital, familial and genetic disorders) | 1 | 0
Deafness (Ear and labyrinth disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Ascites (Gastrointestinal disorders) | 0 | 1
Colitis ischaemic (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Ileus (Gastrointestinal disorders) | 1 | 1
Intestinal ischaemia (Gastrointestinal disorders) | 1 | 1
Intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Mesenteric arteriosclerosis (Gastrointestinal disorders) | 0 | 1
Obstructive pancreatitis (Gastrointestinal disorders) | 1 | 0
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Death (General disorders) | 2 | 2
Multiple organ dysfunction syndrome (General disorders) | 1 | 0
Pyrexia (General disorders) | 1 | 0
Sudden cardiac death (General disorders) | 1 | 0
Vascular stent stenosis (General disorders) | 0 | 1
Acute hepatic failure (Hepatobiliary disorders) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 0
Congestive hepatopathy (Hepatobiliary disorders) | 2 | 0
Hepatic cirrhosis (Hepatobiliary disorders) | 1 | 0
Hepatotoxicity (Hepatobiliary disorders) | 0 | 1
Bacterial infection (Infections and infestations) | 1 | 0
COVID-19 (Infections and infestations) | 3 | 1
COVID-19 pneumonia (Infections and infestations) | 2 | 1
Erysipelas (Infections and infestations) | 0 | 1
Hepatitis A (Infections and infestations) | 1 | 0
Infection (Infections and infestations) | 1 | 0
Infectious pleural effusion (Infections and infestations) | 0 | 1
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 1 | 0
Intervertebral discitis (Infections and infestations) | 1 | 0
Klebsiella infection (Infections and infestations) | 1 | 0
Pelvic abscess (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 4 | 0
Pulmonary sepsis (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 2 | 0
Septic shock (Infections and infestations) | 1 | 1
Staphylococcal bacteraemia (Infections and infestations) | 1 | 0
Subcutaneous abscess (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 1
Urinary tract infection bacterial (Infections and infestations) | 2 | 0
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1
Dislocation of vertebra (Injury, poisoning and procedural complications) | 1 | 0
Eye injury (Injury, poisoning and procedural complications) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 3
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0
Fibula fracture (Injury, poisoning and procedural complications) | 1 | 0
Head injury (Injury, poisoning and procedural complications) | 0 | 1
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 1
Ligament sprain (Injury, poisoning and procedural complications) | 1 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 1 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 1 | 0
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 1 | 0
Blood creatinine increased (Investigations) | 1 | 1
Blood urea increased (Investigations) | 0 | 1
Blood uric acid increased (Investigations) | 0 | 1
Glomerular filtration rate decreased (Investigations) | 1 | 0
International normalised ratio increased (Investigations) | 1 | 0
Troponin increased (Investigations) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 | 1
Gout (Metabolism and nutrition disorders) | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 2
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0
Metabolic acidosis (Metabolism and nutrition disorders) | 1 | 1
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Carotid artery dissection (Nervous system disorders) | 1 | 0
Carotid artery occlusion (Nervous system disorders) | 1 | 0
Cauda equina syndrome (Nervous system disorders) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 3 | 3
Monoplegia (Nervous system disorders) | 1 | 0
Paraplegia (Nervous system disorders) | 1 | 0
Speech disorder (Nervous system disorders) | 1 | 0
Spinal cord compression (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 0 | 1
Toxic encephalopathy (Nervous system disorders) | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 0 | 1
Delirium (Psychiatric disorders) | 1 | 1
Mental status changes (Psychiatric disorders) | 1 | 1
Suicide attempt (Psychiatric disorders) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 19 | 10
Chronic kidney disease (Renal and urinary disorders) | 3 | 0
Hydronephrosis (Renal and urinary disorders) | 1 | 0
Nephropathy (Renal and urinary disorders) | 1 | 0
Nephrotic syndrome (Renal and urinary disorders) | 1 | 0
Renal artery stenosis (Renal and urinary disorders) | 0 | 1
Renal impairment (Renal and urinary disorders) | 4 | 2
Urinary retention (Renal and urinary disorders) | 0 | 1
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 1 | 1
Extremity necrosis (Vascular disorders) | 0 | 1
Hypertensive crisis (Vascular disorders) | 2 | 0
Hypertensive emergency (Vascular disorders) | 1 | 0
Hypotension (Vascular disorders) | 5 | 2
Hypovolaemic shock (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=264) | 10 mg Empagliflozin (N=260)
Hypotension (Vascular disorders) | 19 | 20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2020-06-04): https://cdn.clinicaltrials.gov/large-docs/51/NCT04157751/Prot_000.pdf
  • Statistical Analysis Plan (2021-03-11): https://cdn.clinicaltrials.gov/large-docs/51/NCT04157751/SAP_001.pdf